CLINICAL TRIAL: NCT02452385
Title: Phase 1 Study of CM082 in Patients With wAMD: Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy
Brief Title: Phase 1 Study of CM082 in Patients With wAMD
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor requirements
Sponsor: AnewPharma (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-OPH-101
Record Dates: First submitted 2015-03-10; First posted 2015-05-22 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — vorolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CM082 tablet (Experimental): Escalating dose of CM082 tablet starting at 25mg once a day
  Interventions: Drug: CM082 tablet

INTERVENTIONS:
Drug: CM082 tablet — CM082 tablets taken orally
  Other Names: X-82

SUMMARY:
This is a Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CM082 tablets in Chinese Patients With wAMD.

DETAILED DESCRIPTION:
This is a Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CM082 tablets in Chinese Patients With wAMD. Patients will receive one of four doses for up to four weeks. Single/multiple dose pharmacokinetics in these patients will be studied. At the end of four weeks, investigator will evaluate safety and tolerability and decide whether to continue treatment for a total of six months to further evaluate safety and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Active choroidal neovascularization (CNV) associated with AMD, as evidenced on fluorescein angiography (FA) and OCT.
* Patients with either no previous anti-VEGF therapy or prior anti-VEGF therapy with evidence of response to treatment and the need for additional treatment.
* Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA 20/40 to 20/320 in the study eye(s).
* Adequate bone marrow, hepatic, and renal functions.
* Willing and able to provide written informed consent, comply with the investigational study protocol and return for all study visits.

Exclusion Criteria:

* Patients with Polypoidal Choroidal Vasculopathy (PCV) as evidenced on Indocyanine Green Angiography (ICG).
* Previous treatment with photodynamic therapy (PDT), external beam radiation, subfoveal focal laser photocoagulation, submacular surgery, or transpupillary thermotherapy.
* CNV due to causes other than AMD, including ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia.
* Geographic atrophy involving the foveal center in the study eye.
* Any retinal vascular disease or retinal degeneration other than AMD in the study eye.
* Any significant disease in the study eye that could compromise best-corrected visual acuity.
* Cataract surgery in the study eye within three months of screening.
* Trabeculectomy or aqueous shunt or valve in the study eye.
* Use of any investigational agent or participation in any other clinical trial of an investigational agent or investigational therapy within thirty (30) days of baseline.
* Females of child bearing potential that are pregnant or not using medically acceptable contraception; males unwilling to take adequate contraceptive measures.
* Serious allergy to or prior significant adverse reaction to fluorescein.
* Undiagnosed acute illness first observed during screening or between screening and baseline, or severe concurrent medical conditions that, in the investigators judgment, represent a safety concern.
* Severe cardiac disease, symptomatic congestive heart failure, unstable angina, acute coronary syndrome, myocardial infarction or coronary artery revascularization, or arterial thrombosis within 12 months of start of study drug, inadequately controlled hypertension, or ventricular tachyarrhythmias requiring ongoing treatment.
* QTc ≥450 msec or subjects with a history of risk factors for Torsades de Pointes.
* Stroke or transient ischemic attack within 12 months of trial entry.
* Clinically significant impaired renal or hepatic function.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of CM082.
* Serious active infection, other serious medical condition or any other condition that would impair the ability of the subject to administer the investigational drug or to adhere to the study protocol requirements.
* Presence of any condition which, in the judgment of the investigator, would prevent the subject from completing the study.
* Need to take any medicine that is a strong inhibitor or inducer of CYP3A4.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | six months
  Incidence of the adverse event after treatment

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of CM082 | four weeks
  Single/multiple dose pharmacokinetics in Chinese wAMD patients
Change in best corrected visual acuity (BCVA) (in number of letters) | six months
  Change from baseline in mean BCVA (ETDRS)
Change in Central Retinal Thickness | six months
  Change from baseline in mean central retinal thickness (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, MD, Principal Investigator — West China Hospital
Locations (6):
- China (6):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital，Capital Medical University, Beijing, Beijing Municipality
  - The First People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang